CLINICAL TRIAL: NCT04173455
Title: Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of Bruton Tyrosine Kinase (BTK) Inhibitor HZ-A-018 in Patients With B-Cell Lymphoma
Brief Title: Study of the Safety, Tolerability and Pharmacokinetics of HZ-A-018 in Patients With B Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Hangzhou HeZheng Pharmaceutical Co., Ltd (Unknown)
Responsible Party: Principal Investigator, shentu jianzhong, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZ-A-018-001
Record Dates: First submitted 2019-11-14; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HZ-A-018 (Experimental): In the dose-escalation part, the "3+3" design will be applied. If the subject does not have a DLT during the first 28-day cycle, those who with stable or remission of disease may continue to receive treatment until disease progression, intolerable toxicity or the subject no longer benefits.
  In the dose-expansion part, HZ-A-018 will be administered for several 28-day cycles until disease progression, intolerable toxicity or the subject no longer benefits.
  Interventions: Drug: HZ-A-018

INTERVENTIONS:
Drug: HZ-A-018 — In the dose-escalation part, subjects will be assigned to five cohorts with increaing dose level to determine DLT and MTD during the first 28-day cycle.
  In the expansion part, subjects will be assigned to two fixed dose corhort.

SUMMARY:
The purpose of this study is to establish the safety, tolerability, pharmacokinetics and RP2D (Recommended Phase II Dose) of orally administered HZ-A-018 in patients with B cell lymphoma who have at least failed or relapsed after first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between 18 and 75 years old, voluntarily signed a informed consent.
* Body weight ≥ 45 kg.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0~1.
* Life expectancy (in the opinion of the investigator) of ≥ 4 months.
* Patients with histologically or cytologically confirmed mature B-cell lymphoma according to 2017 WHO (World Health Organization) classification, including chronic lymphocytic leukemia/ small lymphocytic lymphoma (CLL/SLL), mantle cell lymphoma (MCL), follicular lymphoma (FL), marginal zone lymphoma (MZL), Waldenström's Macroglobulinemia (WM) and diffuse large B-cell lymphoma (DLBCL); previous treatment for DLBCL patients must include Rituxan (CD20 monoclonal antibody) and anthracyclines-based therapy and meet one of the following criteria: 1）complete response was not achieved after previous second line therapy; 2) disease progression occurred during any of previous treatment; 3) the duration of stable disease was ≤ 6 months; 4) Disease progression or recurrence occurred within 12 months after autologous hematopoietic stem cell transplantation; CLL and other indolent B-cell NHL patients must meet one of the following criteria: at least failure to respond to first line therapy (SD or PD after treatment with Rituxan-based and alkylating agents or anthracyclines therapy), any response (CR or PR) and progression after stable disease.
* Measurable disease for SLL, MCL, FL, DLBCL and MZL: lymph node lesions>1.5 cm diameter in at least one dimension or any of external node lesions >1.0 cm diameter in at least one dimension; for CLL, peripheral blood monoclonal lymphocytes ≥ 5.0×109/L; for WM, IgM﹥2×ULN (upper limit of normal).
* Any non-hematologic toxicity associated with prior treatment should recover to grade ≤ 1 (according to NCI CTCAE version 5.0).
* Adequate hematological function (no blood transfusion, no use of G-CSF (G-Colony stimulating factor) and no drug correction within 14 days of screening): absolute neutrophil count (ANC) ≥ 0.75 × 109 /L (≥ 0.5×109/L if presence of bone marrow infiltration); platelet count ≥ 50 × 109/L; Hgb ≥ 8.0 g/dL (≥7.0 g/dL if presence of bone marrow infiltration for WM and CLL).
* Adequate renal function: serum creatinine ≤ 1.5 × ULN or estimated creatinine clearance ≥ 60 mL/min (Male: Cr (mL/min) = (140- age) × weight (kg) /72× serum creatinine concentration (mg/dl); Female: Cr (ml/min) = (140- age) × weight (kg) /85× serum creatinine concentration (mg/dl)).
* Adequate liver function: total serum bilirubin ≤ 1.5 x ULN (≤3.0×ULN if presence of liver metastasis); AST and ALT ≤ 2.5 x ULN (≤5.0×ULN if presence of liver metastasis).
* Female of childbearing age and males subjects with fertility must practice at least one of the following effective contraception methods throughout the study and within 90 days of discontinuing study drug: total abstinence from sexual intercourse, physical contraception, or hormonal contraceptive initiated at least 3 months prior to first dose of study drug.
* Male subjects must not donate sperm from initial study drug administration, until 90 days after drug discontinuation.
* Ability to swallow oral capsules without difficulty.
* Willing to follow visit schedules, drug administration schedules, laboratory tests and other test procedures.

Exclusion Criteria:

* Prior BTK inhibitor treatment.
* Infiltration of CNS (central nervous system) by lymphoma.
* Prior organ transplantation or allogeneic hematopoietic stem cell transplantation.
* History of other active malignancies, with exception of basal cell carcinoma of skin, squamous cell carcinoma of skin, cervical carcinoma in situ, or other carcinoma in situ with curative therapy and no recurrence within 5 years.
* Uncontrolled systemic infection or infection requiring intravenously anti-microbial therapy.
* Major surgery or severe trauma within 4 weeks before signing the informed consent.
* Any of the following conditions occurred within the past 6 months: significant cardiac diseases, such as congestive heart failure (NYHA III or IV heart failure), myocardial infarction, and unstable angina pectoris; significant ECG abnormalities, such as atrial fibrillation of any grade, grade II atrioventricular block or grade III atrioventricular block or QTc (F) > 470 msec (female) or > 450 msec (male); other arrhythmias that require treatment.
* Active renal, neurological/psychiatric, liver or endocrine disease, in the opinion of the investigator, would adversely impact on his/her participating in the study.
* Inability to comply with study procedures.
* Stroke or cerebral hemorrhage occurred within 6 months prior to the first dose of the study drug.
* Uncontrolled hypertension, in the opinion of the investigator.
* Previous or active pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, etc.
* Active hepatitis B or C infection (HBV: HBV-DNA ≥1000 IU/mL; hcv: HCV RNA positive with abnormal liver function) or human immunodeficiency virus (HIV) infection or syphilis.
* Active enteritidis , chronic diarrhea, known diverticulosis, or prior gastrectomy or gastric banding, or other conditions that affect absorption.
* Concurrent use of a strong CYP3A4/5 inhibitor (ketoconazole, itraconazole, voriconazole, posaconazole, talimycin, and clarithromycin) or inducers (carbamazepine, rifampicin, phenytoin sodium, etc.) during the study.
* Concurrent use of warfarin or vitamin K antagonists or anticoagulation therapies, or having bleeding tendency or coagulation disorder, within 4 weeks prior to signing the informed consent or during the study.
* Treatment with anti-tumor therapy (including chemotherapy, radiotherapy, immunotherapy, targeted therapy, traditional Chinese medicine or other clinical research therapy) within 4 weeks prior to signing the informed consent; anti-tumor treatment with steroid hormone (dose equivalent to prednisone > 20 mg) within 7 days prior to signing the informed consent.
* Pregnant, breast-feeding or intending to have children with their partners during the study and within 3 months after discontinuation of the study.
* Participating in another clinical trial and taking the drug within 4 weeks prior to signing the informed consent.
* In the opinion of the investigator, other factors that may cause subjects to be forced to terminate the study, such as other serious diseases, serious laboratory abnormalities, and other factors that may affect subjects' safety or test data and blood sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity assessment for each patient | At the end of the first 28 day cycle
  The "3+3" design will be applied in the dose-escalation part.
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 28 days)
  The "3+3" design will be applied in the dose-escalation part.
Adverse events (AEs) | Up to 2 years
  Adverse events at each visit with the NCI CTCAE v5.0 used as a guide for the grading of severity.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | At the end of Cycle 1 (each cycle is 28 days)
Time to reach maximum plasma concentration (Tmax) | At the end of Cycle 1 (each cycle is 28 days)
Area under the plasma concentration-time curve from time zero to t (AUC0~t) | At the end of Cycle 1 (each cycle is 28 days)
Area under the plasma concentration-time curve from time zero to infinity (AUC0~∞) | At the end of Cycle 1 (each cycle is 28 days)
Elimination half-life (t1/2) | At the end of Cycle 1 (each cycle is 28 days)
BTK (Brutons tyrosine kinase) occupancy in PBMCs(peripheral blood mononuclear cells) | At the end of Cycle 1 (each cycle is 28 days)
Objective response rate (ORR) | Up to 2 years
  The proportion of CR (complete response) and PR (partial response).
Duration of response (DOR) | Up to 2 years
  Duration of response is defined as the time from the date of first occurrence of CR (complete response) or PR (partial response) to the date of the first documented PD (progressive disease) or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Shentu, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No